CLINICAL TRIAL: NCT06993597
Title: Development of Robust Corneal Biomechanical Biomarkers for Glaucoma Using Brillouin Microscopy
Brief Title: Study of Corneal Biomechanics in Glaucoma Patients Using Brillouin Microscopy
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HP-00110432; R21EY035483 (NIH)
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma
Keywords: glaucoma; cornea; biomechanics
MeSH Terms: conditions — Glaucoma; Corneal Diseases | interventions — Latanoprost; Bimatoprost; Adrenergic beta-Antagonists; Timolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Normal Tension Glaucoma: Newly diagnosed, treatment-naïve subjects with normal tension glaucoma. Brillouin imaging will be performed at baseline, and in a subset receiving IOP-lowering therapy, additional imaging will be performed at 3 and 6 weeks.
  Interventions: Drug: Prostaglandin Analogue -Containing IOP-Lowering Therapy; Drug: Beta Blocker; Device: Brillouin Microscopy
- High Tension Glaucoma: Newly diagnosed, treatment-naïve subjects with high tension glaucoma. Brillouin imaging will be performed at baseline, and in a subset receiving IOP-lowering therapy, additional imaging will be performed at 3 and 6 weeks.
  Interventions: Drug: Prostaglandin Analogue -Containing IOP-Lowering Therapy; Drug: Beta Blocker; Device: Brillouin Microscopy
- Control: Age-matched healthy control subjects with no history of glaucoma or IOP-lowering therapy. Brillouin imaging will be performed at a single time point for cross-sectional comparison.
  Interventions: Device: Brillouin Microscopy

INTERVENTIONS:
Drug: Prostaglandin Analogue -Containing IOP-Lowering Therapy — Subjects with glaucoma may be prescribed prostaglandin analogs as part of their clinical care. This group will be observed longitudinally to assess changes in corneal biomechanics.
  Other Names: Latanoprost; Travaprost; Bimatoprost
  Groups: High Tension Glaucoma; Normal Tension Glaucoma
Drug: Beta Blocker — Subjects with glaucoma may be prescribed topical beta blockers as part of their clinical care. This group will be observed longitudinally to assess changes in corneal biomechanics.
  Other Names: Timolol
  Groups: High Tension Glaucoma; Normal Tension Glaucoma
Device: Brillouin Microscopy — Brillouin microscopy is a non-contact optical imaging method used to assess the biomechanical properties of the cornea in vivo with three-dimensional resolution. It will be used to evaluate corneal stiffness in all study subjects.
  Other Names: Brillouin Imaging

SUMMARY:
This pilot study evaluates the biomechanical properties of the cornea in glaucoma patients using Brillouin microscopy, a non-contact imaging technique. The study aims to compare corneal stiffness between patients with normal-tension glaucoma, high-tension glaucoma, and healthy controls, and to assess changes in corneal biomechanics following intraocular pressure (IOP)-lowering treatment. The goal is to determine whether Brillouin-derived biomechanical measurements can serve as biomarkers for glaucoma risk and progression.

DETAILED DESCRIPTION:
This study explores the biomechanical properties of the cornea in patients with glaucoma using a novel, non-contact imaging technique called Brillouin microscopy. The technology allows in vivo assessment of tissue stiffness without physical perturbation, potentially offering new insights into glaucoma risk and response to therapy.

The study includes two parts: a cross-sectional comparison between patients with normal- and high-tension glaucoma and healthy controls, and a longitudinal analysis of biomechanical changes following IOP-lowering treatment with either prostaglandin analogs or beta blockers.

The goal is to determine whether corneal biomechanics can serve as a biomarker for glaucoma susceptibility and progression, and to evaluate the feasibility of integrating Brillouin imaging into clinical glaucoma care.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 years or older

Diagnosis of primary open angle glaucoma (POAG) or no history of glaucoma (for controls)

Open angle on gonioscopy (Shaffer grade 3 or 4)

Best-corrected visual acuity of 20/25 or better

Refractive error between +3.00 and -5.00 diopters

No prior use of topical glaucoma medications

Diagnosis of:

High Tension Glaucoma (IOP ≥ 22 mmHg on 3 visits)

Normal Tension Glaucoma (IOP ≤ 21 mmHg on 3 visits)

OR age-matched control with normal optic nerve and visual fields

Exclusion Criteria:

Corneal abnormalities or conditions interfering with Brillouin or applanation tonometry

Retinal diseases affecting RNFL (e.g., macular traction)

History of ocular surgery or laser

Diagnosis of diabetes

History of uveitis

History of prolonged steroid use

Neurodegenerative or systemic diseases (e.g., multiple sclerosis, Alzheimer's, Parkinson's, schizophrenia)

Unreliable visual fields

Contraindications to beta blockers (e.g., bradycardia, severe pulmonary disease)

Moderate to severe glaucoma (per Hodapp-Anderson-Parrish criteria)

History of contact lens use

Low blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 18 years and older with newly diagnosed, treatment-naïve primary open angle glaucoma (POAG), including both normal tension glaucoma (NTG) and high tension glaucoma (HTG), as well as age-matched healthy control subjects. Subjects must meet strict ophthalmic inclusion criteria and will be recruited from the University of Maryland Department of Ophthalmology and Visual Sciences and affiliated clinics. Exclusion criteria include significant ocular comorbidities, prior ocular surgery, systemic diseases that affect the eye, or prior glaucoma therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Corneal Biomechanical Modulus | Baseline, 3 weeks, and 6 weeks
  Brillouin microscopy will be used to measure the corneal modulus of elasticity. The primary outcome is the change in corneal stiffness (Brillouin shift in MHz) across time points in subjects treated with prostaglandin analogs versus beta blockers, and between groups at baseline (NTG, HTG, controls).

CONTACTS AND LOCATIONS:
Overall Officials: Osamah Saeedi, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Summary-level results will be published and made publicly available per NIH policy.